CLINICAL TRIAL: NCT05203211
Title: Use of Testicular Spermatozoa in Non-azoospermic Patients: Retrospective Analysis of a Single Center Experience.
Brief Title: Use of Testicular Spermatozoa in Non-azoospermic Patients
Acronym: NAZOSPERM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: XXX/2022
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men who have undergone icsi from ejaculated semen
- Men who have undergone icsi from testicular sperm
  Interventions: Procedure: Testicular sperm extraction (TESE)

INTERVENTIONS:
Procedure: Testicular sperm extraction (TESE) — During the procedure, the testis is exposed through a small incision and one or more biopsies are taken blindly. A vertical incision is made in the median raphe, skin, dartos and tunica vaginalis to expose tunica albuginea. The tunica albuginea is incised for about 4 mm at upper pole near the head of epididymis.
  Groups: Men who have undergone icsi from testicular sperm

SUMMARY:
Use of testicular spermatozoa in non-azoospermic patients.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the characteristics of couples whose male partner is offered TESE after the failure of previous ICSI technique performed with ejaculated semen. All couples in a third-level University affiliated centre, between January 2010 and January 2020, whose male partner were diagnosed with any type of oligospermia and underwent TESE after ICSI from ejaculated semen, were included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergone testiscular sperm extraction (TESE) after failure of ICSI with the use of ejaculated sperm

Exclusion Criteria:

* Female age >40 yo

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: All couples in a third-level University affiliated centre, between January 2010 and January 2020, whose male partner were diagnosed with any type of oligospermia and underwent TESE after ICSI from ejaculated semen, were included in the analysis.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-02 (Estimated)

PRIMARY OUTCOMES:
fertilization rate (FR) | 10 years
  Evaluate if there is a higher fertilization rate in male patients undergone TESE

SECONDARY OUTCOMES:
Blastulation rate (BR) | 10 years
  Evaluate if there is a higher blastulation rate in male patients undergone TESE
Miscarriage rate (MR) | 10 years
  Evaluate if there is a lower miscarriage rate in male patients undergone TESE

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozmen B, Caglar GS, Koster F, Schopper B, Diedrich K, Al-Hasani S. Relationship between sperm DNA damage, induced acrosome reaction and viability in ICSI patients. Reprod Biomed Online. 2007 Aug;15(2):208-14. doi: 10.1016/s1472-6483(10)60710-9. PMID 17697499
- [Background] Samplaski MK, Dimitromanolakis A, Lo KC, Grober ED, Mullen B, Garbens A, Jarvi KA. The relationship between sperm viability and DNA fragmentation rates. Reprod Biol Endocrinol. 2015 May 14;13:42. doi: 10.1186/s12958-015-0035-y. PMID 25971317
- [Background] Kendall Rauchfuss LM, Kim T, Bleess JL, Ziegelmann MJ, Shenoy CC. Testicular sperm extraction vs. ejaculated sperm use for nonazoospermic male factor infertility. Fertil Steril. 2021 Oct;116(4):963-970. doi: 10.1016/j.fertnstert.2021.05.087. Epub 2021 Jul 4. PMID 34233843
- [Background] Donoso P, Tournaye H, Devroey P. Which is the best sperm retrieval technique for non-obstructive azoospermia? A systematic review. Hum Reprod Update. 2007 Nov-Dec;13(6):539-49. doi: 10.1093/humupd/dmm029. Epub 2007 Sep 24. PMID 17895238
- [Background] Kang YN, Hsiao YW, Chen CY, Wu CC. Testicular sperm is superior to ejaculated sperm for ICSI in cryptozoospermia: An update systematic review and meta-analysis. Sci Rep. 2018 May 18;8(1):7874. doi: 10.1038/s41598-018-26280-0. PMID 29777145